CLINICAL TRIAL: NCT04060095
Title: Impact of Chronic Treatment by β1-adrenergic Antagonists on Nociceptive-Level (NOL) Index Variation After a Standardized Noxious Stimulus Under General Anesthesia: An Observational Study
Brief Title: Impact of Chronic Treatment by β1-adrenergic Antagonists on Nociceptive-Level (NOL) Index Variation After a Standardized Noxious Stimulus Under General Anesthesia
Acronym: BetaNOL
Status: Completed | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Professor Anesthesiology and Pain Medicine, Ciusss de L'Est de l'Île de Montréal
Other Study IDs: 2020-1946
Record Dates: First submitted 2019-07-16; First posted 2019-08-16 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Nociception During Anesthesia in Patients Taking β1-adrenergic Antagonist Chronic Treatment
Keywords: NOL index, anesthesia, β1-adrenergic antagonist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- β1-adrenergic antagonists: Patients who have been treated for more than 3 months with β1-adrenergic antagonists
  Interventions: Procedure: standardized noxious stimulus under general anesthesia.

INTERVENTIONS:
Procedure: standardized noxious stimulus under general anesthesia. — 50 adult patients undergoing general anesthesia for any types of surgery and who have been chronically treated with β1-adrenergic antagonists for at least three months. .Induction of anesthesia will be standardized.
  At least 10 min after the post-intubation decrease of the remifentanil infusion rate, the OR team will stop any physical contact/stimulation of the patient allowing at least 3-minutes.
  At this point, the standardized electrical (tetanic) stimulation will be applied on the area of the ulnar nerve at the wrist level, at a frequency of 100 Hz and a current of 70 mA for a duration of 30 seconds, followed by 3 minutes of observation period without any other stimulation of the patient by the anesthesia or the surgical team. At the end of the observation period, the study is discontinued and the anesthesia will be conducted at the discretion of the anesthesiologist in charge of the patient.

SUMMARY:
The aim of the present study is to investigate the effect of chronic treatment with β1-adrenergic antagonist on the NOL index variation, the heart rate variation and the mean blood pressure variation after a standardized noxious stimulus.

DETAILED DESCRIPTION:
Hypothesis: We hypothesize that the NOL values variations obtained in response to a standardized noxious stimulus under general anesthesia in a group of patients chronically treated with β1-adrenergic antagonists, will be similar to the NOL values variations previously obtained in response to a similar standardized noxious stimulus and previously reported in a group of patients without any β1-adrenergic antagonist.

Background: The Pain Monitoring Device (PMD200TM) monitor (Medasense Biometrics Ltd., Ramat Gan, Israel) uses the Nociception Level (NOL) index, a multiple parameter-derived index that has recently shown a good sensitivity and specificity to detect noxious stimuli. The NOL index variations of the latest version of the PMD200TM has shown better sensitivity and specificity to detect standardized noxious stimulus than heart rate or blood pressure variation in a population without any β1-adrenergic antagonist treatment. β1-adrenergic antagonist treatment was so far a limitation to the use of the NOL index. Indeed, β1-adrenergic antagonists have a depressive action on the heart rate, including limitation of the heart rate variability after a noxious stimulus. Because heart rate and its variability are parameters which are part of the parameters combined to build the NOL index, chronic treatment with β1-adrenergic antagonist could alter the ability of the NOL index to detect noxious stimulus. However, Edry R. (Edry R, 2017) assessed the impact of chronic treatment with β1-adrenergic antagonist on NOL index variation after noxious stimuli in a pilot study (9 patients under chronic treatment with β1-adrenergic antagonist and under general anesthesia) and didn't show any influence of this treatment on the NOL index variation. But this study was not large enough and did not fully answered the question whether chronic treatment with β1-adrenergic antagonist might impact NOL ability to detect precise and standardized stimulus and to compare the results to those in patients without this type of chronic medication.

Objectives:

Primary objective:

To explore the NOL variation in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to standardized noxious stimulus under general anesthesia.

Secondary objectives:

Secondary outcome [1] To explore the heart rate variation and the mean blood pressure variation in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to standardized noxious stimulus under general anesthesia.

Secondary outcome [2] To compare the heart rate variation and the mean blood pressure variation in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to standardized noxious stimulus under general anesthesia to a control group of patients without any β1-adrenergic antagonist chronic treatment; results gathered from a previous study (Renaud-Roy E, 2019), exposed to the same noxious stimulus and under the same anesthesia conditions.

Secondary outcome [3] To explore the ability of the NOL index, the heart rate and the mean blood pressure to discriminate between noxious and non-noxious states in a group of patients with β1-adrenergic antagonist chronic treatment submitted to standardized noxious stimulus under general anesthesia. To determine sensitivity and specificity (ROC curve and AUC of ROC) for each parameter: HR, MAP, NOL index.

Secondary outcome [4] To evaluate the NOL index, the heart rate and the mean blood pressure variations after tracheal intubation in patients with β1-adrenergic antagonist chronic treatment.

Methods:

Adult patients undergoing general anesthesia for any types of surgery and who have been chronically treated with β1-adrenergic antagonists for at least three months prior to surgery will be enrolled to reach a total of patients with full analysis of data of n=25. All patients will be consented prior to the surgery. Induction of anesthesia will be standardized for all patients and based on their adjusted body weight calculated before induction, with: IV midazolam (0.02mg/kg), IV propofol (1.5-2mg.kg-1), IV remifentanil (1mcg.kg-1 followed by a continuous infusion of 0.05 µg.kg-1.min-1), IV rocuronium (0.6 to 1mg.kg-1). Depth of anesthesia with desflurane will be maintained and monitored with the BIS index kept between 40 and 60. Intubation will be performed 3 minutes after the intravenous administration of the propofol, remifentanil and rocuronium boluses. The end of the bolus of remifentanil (given 1mcg/kg; adjusted body weight) will be the start of the 3 min period to wait before proceeding with the tracheal intubation. Three minutes after intubation, the remifentanil infusion will be decreased to 0.005 µg.kg-1.min-1 to reduce the risk of developing hypotensive events and to prepare the patient for the standardized noxious stimulus of the study protocol realized under very low doses of opioids under desflurane hypnosis with BIS 40-60.

At least 10 min after the post-intubation decrease of the remifentanil infusion rate, the OR team will stop any physical contact/stimulation of the patient allowing at least a 3-minutes rest period under stable anesthesia. Baseline mean arterial blood pressure (MAP) and heart rate (HR) will be defined for the rest of the study as the mean of 3 measures in the 3 minutes during this "no pain - no touching" evaluation period to get baselines values of all the study parameters. If necessary, phenylephrine will be given to keep a MAP > 65 mmHg.

At this point, the standardized electrical (tetanic) stimulation will be applied on the area of the ulnar nerve at the wrist level, at a frequency of 100 Hz and a current of 70 mA for a duration of 30 seconds, followed by 3 minutes of observation period without any other stimulation of the patient by the anesthesia or the surgical team (EZstimII, Model ES400, Life-Tech, Stafford, Tx, USA). At the end of the observation period, the study is discontinued and the anesthesia will be conducted at the discretion of the anesthesiologist in charge of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age > 18 years
2. ASA I-III
3. Adult patients scheduled to undergo elective surgery under general anesthesia
4. Patients chronically treated with β1-adrenergic antagonists for at least three months prior to surgery
5. Patient able to consent in the language of the including center

Exclusion Criteria:

1. Use of any type of anesthesia (neuraxial, epidural or local regional anesthesia) without general anesthesia
2. Patients with non-regular sinus cardiac rhythm, implanted pacemakers, prescribed antimuscarinic agents, α2-adrenergic agonists, and antiarrhythmic agents others than β1-adrenergic antagonists
3. Emergent surgery
4. Pregnancy/lactation. Pregnancy test will be performed in all women of child bearing age
5. BMI > 40 kg/m2
6. Preoperative hemodynamic disturbance
7. Central nervous system disorder (neurologic/head trauma/uncontrolled epileptic seizures)
8. Peripheric nervous system disorder (troubles of the peripheric nervous conduction, diabetic neuropathy)
9. Pre-operative chronic opioid use or chronic pain, equivalent to oxycodone 20mg per oral, per day for more than 6 weeks
10. Chronic use of psychoactive drugs within 90 days prior to surgery
11. Medical conditions qualifying for ASA III or IV:

    1. Untreated or persistent peripheral or central cardiovascular disease
    2. Severe pulmonary disease e.g. COPD gold 4, FEV< 1.0l/s, or (evidence of) elevated paCO2 > 6.0 kPa
    3. Significant hepatic disease with increased bilirubin, INR or low albumin
    4. History of severe cardiac arrhythmia eg. Chronic atrial fibrillation.
    5. Active pacemaker or defibrillator
12. Allergy or intolerance to any of the study drugs
13. Cardiac arrhythmia during the period of the study
14. Unexpected difficult airway requesting excessive, possibly painful airway manipulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment of a total of 25 adult patients undergoing general anesthesia for elective surgery (full data analysis available for 25 patients; inclusion until this n is reached). This number was determined on two previous studies conducted at Maisonneuve-Rosemont on the NOL index reactivity to the same stimulus and under the same anesthesia conditions and published in 2018 (Stockle PA et al. Minerva Anestesiologica) and 2019 (Renaud-Roy et al. CJA) from which we got full data from 25 patients who were not chronically treated by β1-adrenergic antagonists. We will compare this previous cohort to the new prospective cohort of patients chronically treated with β1-adrenergic antagonists.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
NOL variation (NOL is an index without unit) before and after stimulation (delta NOL), no unit, varies from 0-100 | Intraoperative, during anesthesia
  To explore the NOL variation between NOL average values before tetanic stimulation at the forearm level, and peak of NOL after stimulation (peak will be considered as an average values of 5 values around the maximal value of NOL, as the definition already used in previous studies) in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to standardized noxious stimulus under general anesthesia.

SECONDARY OUTCOMES:
NOL variation (NOL is an index without unit) before and after tracheal intubation (delta NOL), no unit, varies from 0-100 | Intraoperative, during anesthesia
  To explore the NOL variation between NOL average values before tracheal intubation, and peak of NOL after intubation (peak will be considered as an average values of 5 values around the maximal value of NOL, as the definition already used in previous studies) in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to intubation under general anesthesia.
Heart Rate variation before and after tetanic stimulation (delta heart rate), in beats per minute | Intraoperative, during anesthesia
  To explore the Heart Rate variation between heart rate average values before tetanic stimulation at the forearm level, and peak of heart rate after stimulation (peak will be considered as an average values of 5 values around the maximal value of heart rate, as the definition already used in previous studies) in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to standardized noxious stimulus under general anesthesia.
Heart Rate variation before and after intubation (delta heart rate), in beats per minute | Intraoperative, during anesthesia
  To explore the Heart Rate variation between heart rate average values before tracheal intubation, and peak of heart rate after tracheal intubation (peak will be considered as an average values of 5 values around the maximal value of heart rate, as the definition already used in previous studies) in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to intubation under general anesthesia.
Mean blood pressure variation before and after stimulation (delta mean blood pressure), in mmHg | Intraoperative, during anesthesia
  To explore the Mean Blood Pressure variation between Mean Blood Pressure average values before tetanic stimulation at the forearm level, and peak of Mean Blood Pressure after stimulation (peak will be considered as an average values of 5 values around the maximal value of Mean Blood Pressure, as the definition already used in previous studies) in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to standardized noxious stimulus under general anesthesia.
Mean blood pressure variation before and after intubation (delta mean blood pressure), in mmHg | Intraoperative, during anesthesia
  To explore the Mean Blood Pressure variation between Mean Blood Pressure average values before tracheal intubation, and peak of Mean Blood Pressure after tracheal intubation (peak will be considered as an average values of 5 values around the maximal value of Mean Blood Pressure, as the definition already used in previous studies) in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to tracheal intubation under general anesthesia.
Bispectral index (BIS) variation before and after stimulation (delta BIS), no unit, varies from 0-100 | Intraoperative, during anesthesia
  To explore the BIS index variation between BIS average values before tetanic stimulation at the forearm level, and peak of BIS after stimulation (peak will be considered as an average values of 5 values around the maximal value of BIS, as the definition already used in previous studies) in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to standardized noxious stimulus under general anesthesia.
Bispectral index (BIS) variation before and after tracheal intubation (delta BIS), no unit, varies from 0-100 | Intraoperative, during anesthesia
  To explore the BIS index variation between BIS average values before tracheal intubation, and peak of BIS after intubation (peak will be considered as an average values of 5 values around the maximal value of BIS, as the definition already used in previous studies) in a group of patients under chronic treatment with β1-adrenergic antagonists submitted to intubation under general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PR Richebé, MD PhD, Principal Investigator — CIUSSS Est de l'ile de Montreal
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montreal, Montreal East, Quebec, Canada